CLINICAL TRIAL: NCT04726800
Title: A Pilot Study Investigating the Feasibility to Perform Prospective Circulating Tumor DNA (ctDNA) Profiling in Patients With Colorectal Cancer
Brief Title: Circulating Tumour DNA (ctDNA) as a Prognostic and Predictive Marker in Colorectal Cancer - a Pilot Study
Acronym: CITCCA
Status: Active, not recruiting | Type: Observational
Sponsor: Anna Martling (Other)
Responsible Party: Sponsor-Investigator, Anna Martling, Professor, Senior Consultant Surgeon, Karolinska Institutet
Organization: Karolinska Institutet (Other)
Other Study IDs: 2019-04884
Record Dates: First submitted 2021-01-26; First posted 2021-01-27 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Colorectal Cancer
Keywords: predictive marker; prognostic marker; ctDNA; colon cancer; rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Participants will be asked to donate 30ml blood before surgery (baseline), after surgery at 4-6 weeks, 3-, 6-, 12- and 24 months postoperatively to measure cell-free DNA (cfDNA) in plasma.
  All biospecimens will be shipped to the biobank at Karolinska Institutet for further processing. DNA will be extracted from tumor tissue and whole blood. Targeted sequencing of tumor tissue and germline DNA will be performed using in solution hybridization-based capture at Clinical Genomics, SciLife Lab, Stockholm. Blood in the CITCCA pilot will be profiled prospectively with a two-week turnover, using the ProBio infrastructure, mimicking a real clinical scenario where minimal residual disease (MRD) information will be available in a condense report format.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In clinical practice, there are currently no biomarkers that can guide colorectal cancer treatment in the primary and curative setting. Improved biomarker-based adjuvant treatments would be of greatest value in order to reduce the risk of relapse. There are reasons to believe that measurements of circulating tumor DNA (ctDNA) in plasma could be used to monitor minimal residual disease after surgery. To address this question, a pilot study was conducted with the purpose to demonstrate the feasibility to perform prospective profiling of ctDNA in a cohort of patients with colorectal cancer stage I-III using the already created Nordic infrastructure for clinical research built up for the ALASCCA trial. If the pilot study proves successful, a large randomised controlled Nordic multicenter study is planned where patients with positive ctDNA 4-6 weeks after radical surgery will be randomised to chemotherapy and/or a biologic agent.

ELIGIBILITY:
Inclusion Criteria:

* Colon or rectal cancer tumor stage I-III planned for radical surgery
* Clean Colonoscopy or Computed Tomography (CT) colon within 3 months preoperatively or postoperatively but before randomization
* Patient able to understand and sign written informed consent

Exclusion Criteria:

* Distant metastases
* Other cancers (excluding colorectal cancer or other skin cancer than melanoma) within 3 years from screening
* Significant medical illness that would interfere with study participation
* Pregnancy or breastfeeding females
* Current participation in another clinical trial that will be in conflict with the present study
* Patients who are unlikely to comply with the protocol (e.g. uncooperative attitude, inability to return for subsequent visits) and/or otherwise considered by the Investigator to be unlikely to complete the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The pilot study will include patients diagnosed with colorectal cancer stage I-III invited to participate in the ALASCCA study.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility and logistics of measuring ctDNA | 2 years
Frequency of positive ctDNA postoperatively in relation to tumour stage and oncological outcome. | 3 years
Frequency of positive ctDNA preoperative converted to negative postoperatively. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Anna Martling, Professor, Principal Investigator — Karolinska Institutet
Locations (8):
- Akershus Univeristy Hospital, Oslo, Norway
- Sweden (7):
  - Sahlgrenska University Hospital, Gothenburg
  - Skaraborg Hospital, Skövde
  - Capio Sankt Göran Hospital, Stockholm
  - Danderyd University Hospital, Stockholm
  - Ersta Hospital, Stockholm
  - Karolinska University Hospital, Stockholm
  - South Hospital, Stockholm